CLINICAL TRIAL: NCT02995824
Title: Effectiveness of Raltegravir-Based Antiretroviral Therapy in HIV-HCV Coinfected Liver Transplant Recipients: Retrospective Analysis in a Prospective National Cohort Study (RAL-LT-HIV)
Brief Title: Effectiveness of Raltegravir-Based Antiretroviral Therapy in HIV-HCV Coinfected Liver Transplant Recipients
Acronym: RAL-LT-HIV
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Miro, Senior Consultant, Infectious Diseases, Hospital Clinic of Barcelona
Other Study IDs: 2008-4248
Record Dates: First submitted 2016-11-27; First posted 2016-12-16 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Liver Transplantation; HIV Infections; Antiretroviral Therapy
Keywords: Liver transplantation; HIV infection; Antiretroviral therapy; Raltegravir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Raltegravir-based antiretroviral therapy — To analyze retrospectively the efficacy and safety of raltegravir plus 2 nucleoside reverse transcriptase inhibitors (NRTI) [lamivudine (3TC) or emtricitabine.(FTC) plus abacavir (ABC) or tenofovir (TDF)] [Group 1] versus other ART regimens including boosted PI or NNRTIs [Group 2] in 271 HIV/HCV-coinfected patients who underwent liver transplantation between 2002 and 2012 and were followed until December 2016.

SUMMARY:
This is a retrospective observational multicenter cohort study based on 271 consecutive HIV-HCV coinfected patients who underwent liver transplantation (LT) between 2002 and 2012 in 23 centers from Spain and who were prospectively followed until January 2016. The main objective of this study is to analyze the effectiveness and safety of 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus Raltegravir (RAL)- based antiretroviral therapy (ART) compared to other antiretroviral regimens in liver transplant (LT) HIV-HCV co-infected recipients. In addition, the investigators want to know the rejection rates in patients taking RAL-based ART in comparison with other ART-regimens and to know the efficacy and safety of direct antiviral agents (DAAs) against HCV in HIV-infected liver transplant recipients taking RAL-based ART.

DETAILED DESCRIPTION:
With the advent of combined antiretroviral therapy (cART), patients infected with human immunodeficiency virus type 1 (HIV) are now living longer and dying of illnesses other than acquired immunodeficiency syndrome.

Although outcome of liver transplantation (LT) in HIV and hepatitis C virus (HCV)-coinfected recipients was poorer than in HIV-negative recipients in the pre-HAART era, more recent evidence has demonstrated comparable results in both populations [Roland ME (2006), Terrault N (2012)]. Currently, LT can be performed safely in selected HIV-1-infected patients [Miro JM (2012)]. However, a number of issues persist regarding patient selection, postoperative management, treatment of post-LT HCV recurrence and interactions between antiretroviral and immunosuppressive agents. A key challenge in the post-transplant period is the management of pharmacokinetic interactions between immunosuppressive and antiretroviral drugs, particularly ritonavir-boosted HIV protease inhibitors (PIs), which involve a higher risk of allograft rejection and drug toxicity [van Maarseveen EM (2012)].

Frequent monitoring of the levels of calcineurin inhibitors (e.g., tacrolimus or cyclosporine A) is necessary when PIs are introduced or withdrawn in HIV-infected SOT recipients, because they are strong CYP450 inhibitors.

Furthermore, the pharmacokinetics of corticosteroids and mTOR inhibitors can be affected by PIs. In contrast, non-nucleoside reverse transcriptase inhibitors (NNRTI), which are also commonly used in HAART regimens, are CYP450 inducers and may decrease serum levels of calcineurin inhibitors, with the result that it is necessary to increase their dose to prevent allograft rejection. Raltegravir (RAL) is the first HIV-1 integrase inhibitor approved for clinical practice [Powderly WG (2010)]. It was shown to be highly effective and well tolerated in phase III clinical trials in multidrug-experienced HIV- infected patients and as initial therapy in treatment-naïve patients [Powderly WG (2010)]. RAL is metabolized primarily in the liver via glucuronidation mediated by the UDP glucuronosyltransferase 1A1 (UGT1A1) isoenzyme, although a small percentage is cleared via the kidneys [Kassahun K (2007), Brainard DM (2011)]. RAL is not a substrate of CYP450 and is neither an inducer nor an inhibitor of the main CYP450 enzymes or P-glycoprotein- mediated transport. A favorable pharmacokinetic profile has been demonstrated in HIV-infected LT recipients co-treated with RAL and calcineurin inhibitors (cyclosporine, tacrolimus), mTOR inhibitors, and corticosteroids [van Maarseveen EM (2012), Tricot L (2009)], indicating that RAL is probably well tolerated and efficacious in HIV-infected SOT recipients [Tricot L (2009)]. Preliminary data at the Hospital Clinic of Barcelona (Spain) also suggest that no clinically relevant PK interactions between RAL and mycophenolic acid (MPA), another widely used immunosuppressant [Miro JM et al. (2011)]. Moreover, RAL has few interactions with the new direct acting agents (DAAs) against hepatitis C that may be used in the post-transplant period in order to treat HCV recurrence. The most adequate antiretroviral regimen for HIV-HCV coinfected patients undergoing SOT has not been established. However, switching protease inhibitors or NNRTI-based regimens for a RAL-based regimen at the time of transplantation may be an option to be considered.

Population: Multicenter cohort study based on 271 consecutive HIV-HCV coinfected patients who underwent LT between 2002 and 2012 in 23 centers from Spain who were prospectively followed until January 2016. The study started at 2006 and, for patients who underwent LT between 2002 and 2005, the information was gathered retrospectively and all participants were followed until January 2016.

Antiretroviral treatment was given by the doctors in charge of patients based on their best clinical judgment. Therefore, this is not a clinical trial. Fifty-two percent (142) of HIV-HCV coinfected LT recipients were treated after LT with RAL plus 2 nucleoside reverse transcriptase inhibitors (NRTI) [lamivudine (3TC) or emtricitabine.(FTC) plus abacavir (ABC) or tenofovir (TDF)] [Group 1] and 48% of participants (129) were treated with other ART regimens including boosted PI or NNRTIs [Group 2].

Clinical Outcomes and Measurements:

1. HIV-related: incidence of plasma RNA HIV viral rebound, levels of CD4+ T cells, incidence of opportunistic infections after LT at weeks 48, 96,132 and 240;
2. LT-related: incidence of acute or chronic rejection (biopsy-proven), liver re-transplantation or death at weeks 48, 96, 132 and 240.
3. HCV-related: incidence of progression to F3/F4 (diagnosed by liver biopsy or liver elastography), clinical decompensation of liver cirrhosis at weeks 48,96,132 and 240 or plasma RNA HCV recurrence and DAAs-based HCV treatment outcome (12 weeks-sustained virological response [SVR12]);

All outcomes will be compared between Group 1 and Group 2.

The clinical evaluation, the laboratory tests (including cyclosporine and tacrolimus serum levels), the CD4/CD8 subsets and plasma RNA HIV viral load was collected every 12 weeks up to 144 weeks in accordance with routine clinical practice.

* Study start date: 1st January 2017
* Study end date: 31st July 2017
* First Patient in: 1st Jan 2002
* Last patient out: 31st Nov 2012
* Enrollment period already closed 31-12-2011.
* Ongoing active follow-up. Last visit: January 2016.

Planned duration of current analysis: 6 months (3 months: collecting data; 2 months: data management and analysis; 1 month: manuscript preparation).

The simple size was calculated based on the two primary endpoints (incidence of acute or chronic rejection at 48 weeks and death during the whole follow-up period) and preliminary data observed in solid organ transplant HIV-infected recipients at the Hospital Clinic of Barcelona, Spain [Manzardo C et al. (2015)]. Accepting an alpha risk of 0.05 in a two-sided test with 142 subjects in Group 1 and 129 in Group 2, the statistical power for the two primary endpoints will be: 81%, expecting 25% of chronic or acute rejection at 48 weeks in Group 1 and 41% in Group 2; and 98%, expecting 13% of death in Group 1 and 33% in Group 2, at the end of the whole follow-up.

Categorical variables will be expressed as a frequency (percentage). Continuous variables will be expressed as means ± standard deviation or median [interquartile range] according to normal or non-normal distributions. A negative binomial or Poisson regression will be performed to compare the incidence of outcomes in groups of interest. To compare the levels of CD4+ T cells in groups of interest a lineal regression will be performed. All statistical analysis will be carried out using Stata version 13 (StataCorp. 2013. Stata: Release 13. Statistical Software. College Station, TX: StataCorp LP).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients who underwent liver transplantation between 2002 and 2012 in 23 centers from Spain who were prospectively followed until January 2016

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter cohort study based on 271 consecutive HIV-HCV coinfected patients who underwent LT between 2002 and 2012 in 23 centers from Spain who were prospectively followed until January 2016. The study started at 2006 and, for patients who underwent LT between 2002 and 2005, the information was gathered retrospectively and they were followed until January 2016. HIV-HCV coinfected LT recipients were treated after LT, with RAL plus 2 nucleoside reverse transcriptase inhibitors (NRTI) [lamivudine (3TC) or emtricitabine.(FTC) plus abacavir (ABC) or tenofovir (TDF)] [Group 1] or other ART regimens including boosted PI or NNRTIs [Group 2].
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of plasma RNA HIV viral rebound in plasma after liver transplantation | Through study completion, an average of 3 years
  Plasma HIV viral load above 50 copies/mL

SECONDARY OUTCOMES:
CD4+ T cell evolution after liver transplantation | Through study completion, an average of 3 years
  CD4+ T cell count below 100 cells/mm3
Incidence of acute rejection after liver transplantation | Up to 24 weeks
  Biopsy-proven acute rejection (yes or not)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Miro, MD PhD, Principal Investigator — Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roland ME, Barin B, Huprikar S, Murphy B, Hanto DW, Blumberg E, Olthoff K, Simon D, Hardy WD, Beatty G, Stock PG; HIVTR Study Team. Survival in HIV-positive transplant recipients compared with transplant candidates and with HIV-negative controls. AIDS. 2016 Jan 28;30(3):435-44. doi: 10.1097/QAD.0000000000000934. PMID 26765937
- [Background] Terrault NA, Roland ME, Schiano T, Dove L, Wong MT, Poordad F, Ragni MV, Barin B, Simon D, Olthoff KM, Johnson L, Stosor V, Jayaweera D, Fung J, Sherman KE, Subramanian A, Millis JM, Slakey D, Berg CL, Carlson L, Ferrell L, Stablein DM, Odim J, Fox L, Stock PG; Solid Organ Transplantation in HIV: Multi-Site Study Investigators. Outcomes of liver transplant recipients with hepatitis C and human immunodeficiency virus coinfection. Liver Transpl. 2012 Jun;18(6):716-26. doi: 10.1002/lt.23411. PMID 22328294
- [Background] Miro JM, Montejo M, Castells L, Rafecas A, Moreno S, Aguero F, Abradelo M, Miralles P, Torre-Cisneros J, Pedreira JD, Cordero E, de la Rosa G, Moyano B, Moreno A, Perez I, Rimola A; Spanish OLT in HIV-Infected Patients Working Group investigators. Outcome of HCV/HIV-coinfected liver transplant recipients: a prospective and multicenter cohort study. Am J Transplant. 2012 Jul;12(7):1866-76. doi: 10.1111/j.1600-6143.2012.04028.x. Epub 2012 Apr 4. PMID 22471341
- [Background] van Maarseveen EM, Rogers CC, Trofe-Clark J, van Zuilen AD, Mudrikova T. Drug-drug interactions between antiretroviral and immunosuppressive agents in HIV-infected patients after solid organ transplantation: a review. AIDS Patient Care STDS. 2012 Oct;26(10):568-81. doi: 10.1089/apc.2012.0169. PMID 23025916
- [Background] Powderly WG. Integrase inhibitors in the treatment of HIV-1 infection. J Antimicrob Chemother. 2010 Dec;65(12):2485-8. doi: 10.1093/jac/dkq350. Epub 2010 Sep 18. PMID 20852268
- [Background] Kassahun K, McIntosh I, Cui D, Hreniuk D, Merschman S, Lasseter K, Azrolan N, Iwamoto M, Wagner JA, Wenning LA. Metabolism and disposition in humans of raltegravir (MK-0518), an anti-AIDS drug targeting the human immunodeficiency virus 1 integrase enzyme. Drug Metab Dispos. 2007 Sep;35(9):1657-63. doi: 10.1124/dmd.107.016196. Epub 2007 Jun 25. PMID 17591678
- [Background] Brainard DM, Wenning LA, Stone JA, Wagner JA, Iwamoto M. Clinical pharmacology profile of raltegravir, an HIV-1 integrase strand transfer inhibitor. J Clin Pharmacol. 2011 Oct;51(10):1376-402. doi: 10.1177/0091270010387428. Epub 2011 Jan 5. PMID 21209233
- [Background] Tricot L, Teicher E, Peytavin G, Zucman D, Conti F, Calmus Y, Barrou B, Duvivier C, Fontaine C, Welker Y, Billy C, de Truchis P, Delahousse M, Vittecoq D, Salmon-Ceron D. Safety and efficacy of raltegravir in HIV-infected transplant patients cotreated with immunosuppressive drugs. Am J Transplant. 2009 Aug;9(8):1946-52. doi: 10.1111/j.1600-6143.2009.02684.x. Epub 2009 Jun 10. PMID 19519819
- [Background] Miro JM, et al. Combination of Raltegravir (RAL) plus Lamivudine (3TC) or Emtricitabine (FTC) plus Abacavir (ABV) or Tenofovir (TDF) is Safe, Effective and Prevents Pharmacokinetic (PK) Interactions with Immunosuppressive Drugs (IS) in HIV-1-infected Solid Organ Transplant (SOT) Recipients. 18th Conference on Retroviruses and Opportunistic Infections (CROI). Boston, MA. February 27- March 2, 2011. Abstract #644
- [Background] Manzardo C, et al. Raltegravir (RAL) Based Antiretroviral Therapy (ART) in HIV-infected Solid Organ Transplant (SOT) Recipients: a Single Center Experience. 15th EACS Conference. Barcelona, Spain. October 21- 24 2015. Abstract #PE8/68.